CLINICAL TRIAL: NCT02122848
Title: Effects of Bilevel Positive Airway Pressure on Exercise Tolerance in Patients With Decompensated Heart Failure
Brief Title: Exercise Tolerance in Patients With Decompensated Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Sirio-Libanes (Other)
Responsible Party: Principal Investigator, Wellington Yamaguti, Wellington Pereira dos Santos Yamaguti, Hospital Sirio-Libanes
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: hsl 2013-48
Record Dates: First submitted 2014-04-20; First posted 2014-04-25 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Heart Failure
Keywords: Heart failure; Exercise tolerance; Noninvasive ventilation
MeSH Terms: conditions — Heart Failure | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bilevel (Experimental): The intervention will be performed using BiLevel ventilation mode with EPAP=10 cmH2O and a IPAP which manages 6-8ml/kg tidal volume.
  Interventions: Device: BiLevel

INTERVENTIONS:
Device: BiLevel — The intervention will be performed using BiLevel ventilation mode with EPAP=10 cmH2O and a IPAP which manages 6-8ml/kg tidal volume.
  Other Names: BiPAP

SUMMARY:
The purpose of this study is to evaluate the effects of airway bilevel positive pressure on the improvement of exercise tolerance in patients with decompensated heart failure.

DETAILED DESCRIPTION:
Heart failure causes limitation of functional capacity and worsening of exercise tolerance. The airway pressure as adjuvant of cardiac rehabilitation has demonstrated improvement of functional capacity, decrease of respiratory work, increase of oxygenation and pulmonary compliance. Objective: to evaluate the effectiveness of the bilevel positive airway pressure (BILEVEL) in the increase of exercise tolerance in patients with decompensated heart failure. Method: this is a cross-over randomized clinical trial, with individuals who will undergo a submaximal progressive exercise test of the lower limbs with a cycle-ergometer using continuous positive airway pressure (CPAP) and BILEVEL in a random order. Patients will also be evaluated using a health related quality of life questionnaire, pulmonary function test, inspiratory muscle and peripheral muscle strength tests. Hypothesis: The increase in exercise tolerance might be greater during the use of BILEVEL.

ELIGIBILITY:
Inclusion Criteria:

* subjects who has heart failure functional class II or III of New York heart association
* over 18 years
* non-smokers
* without cognitive or motor deficit
* without vasoactive drugs or low doses
* without recent acute myocardial myocardium (<1 year)
* without recent cardiac surgery (<1 year)
* without pulmonary disease
* without bronchodilators

Exclusion Criteria:

* unstable angina
* atrial fibrillation and atrioventricular block third degree
* frequent vomiting
* respiratory instability while collecting data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Endurance time of exercise in cycle ergometer. | 4 days

SECONDARY OUTCOMES:
Dyspnea | 4 days
  Dyspnea will be evaluated by means of the modified Borg scale before and after exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Wellington Yamaguti, Principal Investigator — Hospital Sirio-Libanes
Locations (1):
- Hospitalsiriolibanes, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Moraes IG, Kimoto KM, Fernandes MB, Grams ST, Yamaguti WP. Adjunctive Use of Noninvasive Ventilation During Exercise in Patients With Decompensated Heart Failure. Am J Cardiol. 2017 Feb 1;119(3):423-427. doi: 10.1016/j.amjcard.2016.10.025. Epub 2016 Nov 1. PMID 27939229